CLINICAL TRIAL: NCT00386776
Title: Cybermedicine for the Patient and Physician
Brief Title: Patient Computer Dialog in Primary Care
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Library of Medicine (NLM) (NIH)
Responsible Party: Principal Investigator, Warner Slack, Professor of Medicine, Harvard Medical School, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2004P-000420; R01LM008255-01A1 (NIH)
Record Dates: First submitted 2006-10-11; First posted 2006-10-12 (Estimated); Results first posted 2013-06-10 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2013-06

CONDITIONS: Patient Computer Dialog
Keywords: computers; diagnosis; medical records; physician patient relations; medical history taking; medical informatics applications
MeSH Terms: conditions — Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 'Computer-based medical history (Experimental): A computer-based medical history to take in their homes via the Internet. The history is divided into 24 modules- family history, social history, cardiac history, pulmonary history, and the like.
  Interventions: Other: Computer-based medical history

INTERVENTIONS:
Other: Computer-based medical history — The intervention is a computer-based medical interview, which contains 232 primary questions that are asked of all respondents, and over 6000 frames (questions, explanations, suggestions, recommendations, and words of encouragement) that are available for presentation as determined by the patient's responses and the branching logic of the program.

SUMMARY:
With this clinical study, we hoped to find out if interactive, computer-based medical interviews, when carefully tested and honed and made available to patients in their homes on the Internet, will improve both the efficiency and quality of medical care and be well received and found helpful by patients and their physicians. We developed the computer-based medical interview consisting of over 6000 questions and a corresponding program that provides a concisely written, summary of the patient's responses to the questions in the interview. We then conducted read aloud and test/retest reliability evaluations of the interview and summary programs and determined the programs to be reliable. Results were published in the November 27, 2010 issue of the Journal of the American medical Informatics Association. We also developed, edited, and revised a program that provides a concisely written, summary of the patient's responses to the questions in the interview.

We obtained a grant from the Rx Foundation to conduct clinical trial of our medical history. At the time of the office visit, the summary of the computer-based history of those patients who had completed the interview was available on the doctor's computer screen for the doctor and patient to use together on a voluntary basis. The results of this trial were published in the January 2012 issue of the Journal of the American Informatics Association.

DETAILED DESCRIPTION:
We developed a computer-based medical history for patients to take in their homes via the Internet. The history is divided into 24 modules- family history, social history, cardiac history, pulmonary history, and the like. So far as possible, it is designed to model the comprehensive, inclusive, general medical history traditionally taken, when time permits, by a primary care doctor seeing a patient for the first time. It contains 232 primary questions asked of all patients about the presence or absence of medical problems. Of these, 215 have the preformatted mutually exclusive responses "Yes," "No," "Uncertain (Don't Know, Maybe)," "Don't understand," and "I'd rather not answer;" 10 have other sets of multiple choices, one response permitted; five have multiple choices with more than one response permitted, and two have numerical responses. In addition, more than 6000 questions, explanations, suggestions, and recommendations are available for presentation, as determined by the patient's responses and the branching logic of the program. These questions are available to explore in detail medical problems elicited by one or more of the primary questions. If for example, a patient responds with "Yes" to the question about chest pain, the program branches to multiple qualifying questions about characteristics of the pain, such as onset, location, quality, severity, relationship to exertion, and course. Once we had completed the interview in preliminary form, we made it available to members of our medical advisory board for their criticisms and suggestions. We then conducted a formal read-aloud assessment in which 10 volunteer patients read each primary question aloud to an investigator in attendance and offered their understanding and general assessment of the questions. We revised our program based on comments from the advisory board and the patients

We then conducted a test/retest reliability study of the 215 of the 232 primary questions that have the preformatted, allowable response set of "Yes," "No," "Uncertain (Don't know, Maybe)," "Don't understand," and "I'd rather not answer, the 10 questions that have other response sets with one answer permitted, and the 5 questions with more than one response permitted. Email messages were sent via PatientSite (our patients' portal to their electronic medical record) to inform patients of the study and how to sign on to the informed consent form, and for those that had consented to the study to remind them to take interview for the first and then the second time.)

From randomly selected patients of doctors affiliated with Beth Israel Deaconess Medical Center in Boston, 48 patients took the history twice with intervals between sessions ranging from one to 35 days (mean seven days; median five days). When we analyzed the inconsistency between first and second interviews with which the 48 patients responded to each of the primary questions. We found that the 215 questions with response options of "Yes," "No," "Uncertain," "Don't understand," and "I'd rather not answer" had the lowest incidence (6 percent); the 10 other multiple choice questions with one response permitted had a 13 percent incidence, and the five multiple choice questions with more than one response permitted had a 14 percent incidence. Whenever an inconsistency was detected with the repeat interview, the patient was asked to choose when appropriate from four possible reasons. Reasons chosen were: "clicked on the wrong choice" (23 percent), "not sure about the answer" (23 percent), "medical situation changed" (6 percent), and "didn't understand the question (less than 1 percent). With the remaining 47 percent of the inconsistencies, no reason was given.

We then computed the percentage of agreement for each of the primary questions together with Cohen's Kappa Index of Reliability. Of the 215 "Yes," "No," "Uncertain (Don't know, Maybe)," "Don't understand," and "I'd rather not answer" questions, 96 (45 percent) had kappa values greater than .75 (excellent agreement by the criteria of Landis and Koch, and of these, 38 had kappa values of one (perfect agreement); an additional 24 primary questions (12 percent), to which all patients had made identical responses both times (perfect consistency), had no Kappa values. Sixty-eight of these questions (32 percent) had kappa values between .40 and .75 (fair to good agreement); and 26 (13 percent) had kappa values less than .40 (poor agreement). Of the 27 questions with poor kappa values, 15 had percentages of agreement greater than 90 percent, and we deemed these to be sufficiently reliable within their clinical context to remain unrevised. We selected the 12 questions with poor kappa values and percentages of agreement less than 90 percent for rewording. Of the 15 primary questions with varying sets of responses, half had kappa values in the excellent range and half had kappa values in the fair to good range, and we kept these in place unrevised. Fifteen of the primary questions (7 percent) received a "don't understand" response. Although there was but a single "don't understand" response for each of these questions, we were able to isolate seven with which the possibility of confusion seemed to be evident, and we revised these accordingly.

With the first of the two interviews-with a mean of 545 frames presented and a completion time of 45 to 90 minutes (based on an estimated 7 seconds per frame -the volunteers were for the most part favorable in their assessment of the interview when asked a set of 10, 10-point Likert-scale questions.

These results were published in the November 2010 issue of the Journal of the American Informatics Association.

We also developed, edited, and revised a program that provides a concisely written, summary of the patient's responses to the questions in the interview. This was a formidable project that took considerably longer than we had anticipated. The "phrase" is the basic unit of the summary. Identified by its unique reference number, each phrase contains the words to be generated, the conditions for writing them, and the branching logic that determines the course of the program as it progresses from phrase to phrase. The summary program for the General Medical Interview, which contains over 5,000 phrases, is organized by sections that are related by name and content to their corresponding interview sections. Designed for use by both doctor and patient and available in both electronic and printed form, the summary is presented in a legible but otherwise traditional format.

We were not able to complete the randomized control study at this time due to a couple of factors. First, it took substantially longer than anticipated to develop and evaluate our program in our effort to have a comprehensive, detailed computer-based medical interview that would compare favorably with that of a thoughtful physician. It took us two years to develop, test, and revise the General Medical Interview and far longer than we had anticipated to complete the test-retest reliability study and to develop, test, and revise the summary program. In addition, our medical center's current policy is to obtain a patient's e-mail address only after the patient has had a first visit to the center and only if the patient has been registered in PatientSite after a first visit. Therefore, although we could readily recruit by e-mail our participants for the test-retest study, we were limited to the far more labor-intensive process of telephone recruitment for the randomized, controlled study.

We later obtained a grant from the Rx Foundation us to conduct clinical trial of our newly revised medical history. After completing the medical history the patients were asked to complete an online 10 item 10-point Likert-scale post-history assessment questionnaire. At the time of the office visit, the summary of the computer-based history of those patients who had completed the interview was available on the doctor's computer screen for the doctor and patient to use together on a voluntary basis. At the option of the doctor, the summary could then be edited and incorporated into the patient's online medical record. The day after the visit the patients and the doctors were asked to complete a 10-point Likert-scale questionnaire consisting of six questions that asked about the effect of the medical history and its summary on the quality of the visit from the patient's and the doctor's perspectives, with provision for them to record comments and suggestions for improvement.

The results of this were published in the January 2012 issue of the Journal of the American Informatics Association.

ELIGIBILITY:
Inclusion Criteria:

* Request for an initial appointment with a primary care physician at Beth Israel Deaconess Medical Center who has agreed to participate in the study
* English as first language
* Internet access at home

Exclusion Criteria

* Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2005-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Warner V Slack, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Slack WV, Hicks GP, Reed CE, Van Cura LJ. A computer-based medical-history system. N Engl J Med. 1966 Jan 27;274(4):194-8. doi: 10.1056/NEJM196601272740406. No abstract available. PMID 5902618
- [Background] Bachman JW. The patient-computer interview: a neglected tool that can aid the clinician. Mayo Clin Proc. 2003 Jan;78(1):67-78. doi: 10.4065/78.1.67. PMID 12528879
- [Background] Sands DZ, Halamka JD, Pellaton D. PatientSite: a Web-based clinical communication and health education tool. Proc Annu Conf Health Information Management Systems Society 2001, Chicago, IL (on CD).
- [Background] Slack WV. The computer and the doctor-patient relationship. MD Comput. 1989 Nov-Dec;6(6):320-1. No abstract available. PMID 2607929
- [Background] Slack WV. Patient-Computer Dialogue: A Review. Yearb Med Inform. 2000;(1):71-78. PMID 27699348
- [Background] Slack WV. Cybermedicine: how computing empowers doctors and patients for better health care (revised and updated edition). San Francisco: Jossey-Bass, 2001
- [Background] Forster AJ, Murff HJ, Peterson JF, Gandhi TK, Bates DW. The incidence and severity of adverse events affecting patients after discharge from the hospital. Ann Intern Med. 2003 Feb 4;138(3):161-7. doi: 10.7326/0003-4819-138-3-200302040-00007. PMID 12558354
- [Background] BRODMAN K, ERDMANN AJ Jr, et al. The Cornell medical index; a adjunct to medical interview. J Am Med Assoc. 1949 Jun 11;140(6):530-4. doi: 10.1001/jama.1949.02900410026007. No abstract available. PMID 18144531
- [Background] BRODMAN K, VAN WOERKOM AJ, ERDMANN AJ Jr, GOLDSTEIN LS. Interpretation of symptoms with a data-processing machine. AMA Arch Intern Med. 1959 May;103(5):776-82. doi: 10.1001/archinte.1959.00270050098015. No abstract available. PMID 13636498
- [Background] COLLEN MF, RUBIN L, NEYMAN J, DANTZIG GB, BAER RM, SIEGELAUB AB. AUTOMATED MULTIPHASIC SCREENING AND DIAGNOSIS. Am J Public Health Nations Health. 1964 May;54(5):741-50. doi: 10.2105/ajph.54.5.741. No abstract available. PMID 14153274
- [Background] Slack WV, Van Cura LJ. Computer-based patient interviewing. Postgrad Med. 1968 Apr;43(4):115-20 concl. doi: 10.1080/00325481.1968.11693217. No abstract available. PMID 5689697
- [Background] Slack WV, Van Cura LJ. Computer-based patient interviewing. 1. Postgrad Med. 1968 Mar;43(3):68-74. doi: 10.1080/00325481.1968.11693177. No abstract available. PMID 5650983
- [Background] Peckham BM, Slack WV, Carr WF, Van Cura LJ, Schultz AE. Computerized data collection in the management of uterine cancer. Clin Obstet Gynecol. 1967 Dec;10(4):1003-15. doi: 10.1097/00003081-196712000-00015. No abstract available. PMID 4871715
- [Background] Maultsby MC Jr, Slack WV. A computer-based psychiatry history system. Arch Gen Psychiatry. 1971 Dec;25(6):570-2. doi: 10.1001/archpsyc.1971.01750180090014. No abstract available. PMID 5141376
- [Background] Chun RW, Van Cura LJ, Spencer M, Slack WV. Computer interviewing of patients with epilepsy. Epilepsia. 1976 Dec;17(4):371-5. doi: 10.1111/j.1528-1157.1976.tb04448.x. PMID 1001281
- [Background] Leviton A, Slack WV, Masek B, Bana D, Graham JR. A computerized behavioral assessment for children with headaches. Headache. 1984 Jul;24(2):182-5. doi: 10.1111/j.1526-4610.1984.hed2404182.x. No abstract available. PMID 6400563
- [Background] Bana DS, Leviton A, Swidler C, Slack W, Graham JR. A computer-based headache interview: acceptance by patients and physicians. Headache. 1980 Mar;20(2):85-9. doi: 10.1111/j.1526-4610.1980.hed2002085.x. No abstract available. PMID 7372476
- [Background] Bennett SE, Lawrence RS, Fleischmann KH, Gifford CS, Slack WV. Profile of women practicing breast self-examination. JAMA. 1983 Jan 28;249(4):488-91. PMID 6848849
- [Background] Slack WV, Van Cura LJ. Patient reaction to computer-based medical interviewing. Comput Biomed Res. 1968 May;1(5):527-31. doi: 10.1016/0010-4809(68)90018-9. No abstract available. PMID 5696987
- [Background] Slack WV. A history of computerized medical interviews. MD Comput. 1984;1(5):52-9, 68. No abstract available. PMID 6571302
- [Background] Mayne JG, Weksel W, Sholtz PN. Toward automating the medical history. Mayo Clin Proc. 1968 Jan;43(1):1-25. No abstract available. PMID 5635452
- [Background] Mayne JG, Martin MJ. Computer-aided history acquisition. Med Clin North Am. 1970 Jul;54(4):825-33. No abstract available. PMID 5425111
- [Background] Coombs GJ, Murray WR, Krahn DW. Automated medical histories: factors determining patient performance. Comput Biomed Res. 1970 Apr;3(2):178-81. doi: 10.1016/0010-4809(70)90024-8. No abstract available. PMID 5431936
- [Background] Grossman JH, Barnet GO, McGuire MT, Swedlow DB. Evaluation of computer-acquired patient histories. JAMA. 1971 Feb 22;215(8):1286-91. No abstract available. PMID 5107557
- [Background] Warner HR, Rutherford BD, Houtchens B. A sequential Bayesean approach to history taking and diagnosis. Comput Biomed Res. 1972 Jun;5(3):256-62. doi: 10.1016/0010-4809(72)90087-0. No abstract available. PMID 4555663
- [Background] Stead WW, Heyman A, Thompson HK, Hammond WE. Computer-assisted interview of patients with functional headache. Arch Intern Med. 1972 Jun;129(6):950-5. No abstract available. PMID 4555941
- [Background] Simborg DW, Rikli AE, Hall P. Experimentation in medical history-taking. JAMA. 1969 Nov 24;210(8):1443-5. No abstract available. PMID 5395419
- [Background] Coddington RD, King TL. Automated history taking in child psychiatry. Am J Psychiatry. 1972 Sep;129(3):276-82. doi: 10.1176/ajp.129.3.276. No abstract available. PMID 4559782
- [Background] Gottlieb GL, Beers RF Jr, Bernecker C, Samter M. An approach to automation of medical interviews. Comput Biomed Res. 1972 Apr;5(2):99-107. doi: 10.1016/0010-4809(72)90073-0. No abstract available. PMID 5030841
- [Background] Greist JH, Gustafson DH, Stauss FF, Rowse GL, Laughren TP, Chiles JA. A computer interview for suicide-risk prediction. Am J Psychiatry. 1973 Dec;130(12):1327-32. doi: 10.1176/ajp.130.12.1327. No abstract available. PMID 4585280
- [Background] Rockart JF, McLean ER, Hershberg PI, Bell GO. An automated medical history system. Experience of the Lahey Clinic Foundation with computer-processed medical histories. Arch Intern Med. 1973 Sep;132(3):348-58. doi: 10.1001/archinte.132.3.348. No abstract available. PMID 4593190
- [Background] Schuman SH, Curry HB, Braunstein ML, Schneeweiss R, Jebaily GC, Glazer HM, Cahn JR, Crigler WH. A computer-administered interview on life events: improving patient-doctor communication. J Fam Pract. 1975 Aug;2(4):263-9. PMID 1185132
- [Background] Pauker SG, Gorry GA, Kassirer JP, Schwartz WB. Towards the simulation of clinical cognition. Taking a present illness by computer. Am J Med. 1976 Jun;60(7):981-96. doi: 10.1016/0002-9343(76)90570-2. PMID 779466
- [Background] Lucas RW, Card WI, Knill-Jones RP, Watkinson G, Crean GP. Computer interrogation of patients. Br Med J. 1976 Sep 11;2(6036):623-5. doi: 10.1136/bmj.2.6036.623. PMID 786434
- [Background] Lucas RW, Mullin PJ, Luna CB, McInroy DC. Psychiatrists and a computer as interrogators of patients with alcohol-related illnesses: a comparison. Br J Psychiatry. 1977 Aug;131:160-7. doi: 10.1192/bjp.131.2.160. PMID 334310
- [Background] Lucas RW. A study of patients' attitudes to computer interrogation. Int J Man Machine Studies 1977; 9: 69-86.
- [Background] Greist JH, Klein MH. Computer programs for patients, clinicians, and researchers in psychiatry. In: Sidowski JB, Johnson JH, Williams TA, eds. Technology in mental health care delivery systems. Norwood, Conn.: Ablex, 1980: 161-82.
- [Background] Carr AC, Ghosh A, Ancill RJ. Can a computer take a psychiatric history? Psychol Med. 1983 Feb;13(1):151-8. doi: 10.1017/s0033291700050157. PMID 6844461
- [Background] Carr AC, Ghosh A. Response of phobic patients to direct computer assessment. Br J Psychiatry. 1983 Jan;142:60-5. doi: 10.1192/bjp.142.1.60. PMID 6831131
- [Background] Skinner HA, Allen BA. Does the computer make a difference? Computerized versus face-to-face versus self-report assessment of alcohol, drug, and tobacco use. J Consult Clin Psychol. 1983 Apr;51(2):267-75. doi: 10.1037//0022-006x.51.2.267. No abstract available. PMID 6841771
- [Background] Millstein SG, Irwin CE Jr. Acceptability of computer-acquired sexual histories in adolescent girls. J Pediatr. 1983 Nov;103(5):815-9. doi: 10.1016/s0022-3476(83)80493-4. PMID 6631616
- [Background] Tanser AR, Davies A. Archie: the use of a microcomputer in an allergy clinic. Br J Dis Chest. 1984 Apr;78(2):135-9. PMID 6722016
- [Background] Quaak MJ, Westerman RF, Schouten JA, Hasman A, van Bemmel JH. Patient appreciations of computerized medical interviews. Med Inform (Lond). 1986 Oct-Dec;11(4):339-50. doi: 10.3109/14639238608997657. PMID 3821297
- [Background] Houziaux MO, Lefebvre PJ. Historical and methodological aspects of computer-assisted medical history-taking. Med Inform (Lond). 1986 Apr-Jun;11(2):129-43. doi: 10.3109/14639238609001366. PMID 3526028
- [Background] Lindberg G, Seensalu R, Nilsson LH, Forsell P, Kagar L, Knill-Jones RP. Transferability of a computer system for medical history taking and decision support in dyspepsia. A comparison of indicants for peptic ulcer disease. Scand J Gastroenterol Suppl. 1987;128:190-6. doi: 10.3109/00365528709090990. PMID 3306899
- [Background] Haug PJ, Warner HR, Clayton PD, Schmidt CD, Pearl JE, Farney RJ, Crapo RO, Tocino I, Morrison WJ, Frederick PR. A decision-driven system to collect the patient history. Comput Biomed Res. 1987 Apr;20(2):193-207. doi: 10.1016/0010-4809(87)90045-0. PMID 3595100
- [Background] Pringle M. Using computers to take patient histories. BMJ. 1988 Sep 17;297(6650):697-8. doi: 10.1136/bmj.297.6650.697. No abstract available. PMID 3147730
- [Background] Lutner RE, Roizen MF, Stocking CB, Thisted RA, Kim S, Duke PC, Pompei P, Cassel CK. The automated interview versus the personal interview. Do patient responses to preoperative health questions differ? Anesthesiology. 1991 Sep;75(3):394-400. PMID 1888045
- [Background] Sanders GD, Owens DK, Padian N, Cardinalli AB, Sullivan AN, Nease RF. A computer-based interview to identify HIV risk behaviors and to assess patient preferences for HIV-related health states. Proc Annu Symp Comput Appl Med Care. 1994:20-4. PMID 7949919
- [Background] Hasley S. A comparison of computer-based and personal interviews for the gynecologic history update. Obstet Gynecol. 1995 Apr;85(4):494-8. doi: 10.1016/0029-7844(95)00012-G. PMID 7898822
- [Background] Vitkun SA, Gage JS, Anderson DH 2nd, Williams SA, Halpern-Lewis JG, Poppers PJ. Computerization of the preoperative anesthesia interview. Int J Clin Monit Comput. 1995 May;12(2):71-6. doi: 10.1007/BF01142486. No abstract available. PMID 8847468
- [Background] Kobak KA, Greist JH, Jefferson JW, Katzelnick DJ. Computer-administered clinical rating scales. A review. Psychopharmacology (Berl). 1996 Oct;127(4):291-301. doi: 10.1007/s002130050089. PMID 8923563
- [Background] Taenzer PA, Sauve L, Burgess ED, Milkavich L, Whitmore B. The health interview: automated assessment in a multidisciplinary outpatient hypertension treatment program. MD Comput. 1996 Sep-Oct;13(5):423-6. PMID 8824103
- [Background] Kohlmeier L, Mendez M, McDuffie J, Miller M. Computer-assisted self-interviewing: a multimedia approach to dietary assessment. Am J Clin Nutr. 1997 Apr;65(4 Suppl):1275S-1281S. doi: 10.1093/ajcn/65.4.1275S. PMID 9094933
- [Background] Bock B, Niaura R, Fontes A, Bock F. Acceptability of computer assessments among ethnically diverse, low-income smokers. Am J Health Promot. 1999 May-Jun;13(5):299-304. doi: 10.4278/0890-1171-13.5.299. PMID 10538645
- [Background] Pierce B. The use of instant medical history in a rural clinic. Case study of the use of computers in an Arkansas physician's office. J Ark Med Soc. 2000 May;96(12):444-7. PMID 10846345
- [Background] Rhodes KV, Lauderdale DS, Stocking CB, Howes DS, Roizen MF, Levinson W. Better health while you wait: a controlled trial of a computer-based intervention for screening and health promotion in the emergency department. Ann Emerg Med. 2001 Mar;37(3):284-91. doi: 10.1067/mem.2001.110818. PMID 11223765
- [Background] Locke SE, Kowaloff HB, Hoff RG, Safran C, Popovsky MA, Cotton DJ, Finkelstein DM, Page PL, Slack WV. Computer-based interview for screening blood donors for risk of HIV transmission. JAMA. 1992 Sep 9;268(10):1301-5. PMID 1507376
- [Background] Slack WV. Patient power: a patient oriented value system. In: Jacques JA, ed. Computer diagnosis and diagnostic methods. Proceedings of the Second Conference on the Diagnostic Process held at the University of Michigan. Springfield, IL: Charles C. Thomas, 1972: 3-7.
- [Background] Slack WV. The patient's right to decide. Lancet. 1977 Jul 30;2(8031):240. doi: 10.1016/s0140-6736(77)92849-5. No abstract available. PMID 79024
- [Background] Bloom SM, White RJ, Beckley RF, Slack WV. Converse: a means to write, edit, administer, and summarize computer-based dialogue. Comput Biomed Res. 1978 Apr;11(2):167-75. doi: 10.1016/0010-4809(78)90028-9. No abstract available. PMID 354858
- [Background] Witschi J, Porter D, Vogel S, Buxbaum R, Stare FJ, Slack W. A computer-based dietary counseling system. J Am Diet Assoc. 1976 Oct;69(4):385-90. PMID 956580
- [Background] Slack W, Porter D, Witschi J, Sullivan M, Buxbaum R, Stare FJ. Dietary interviewing by computer. An experimental approach to counseling. J Am Diet Assoc. 1976 Nov;69(5):514-7. PMID 977878
- [Background] Fisher LA, Johnson TS, Porter D, Bleich HL, Slack WV. Collection of a clean voided urine specimen: a comparison among spoken, written, and computer-based instructions. Am J Public Health. 1977 Jul;67(7):640-4. doi: 10.2105/ajph.67.7.640. PMID 327837
- [Background] Slack WV, Safran C, Kowaloff HB, Pearce J, Delbanco TL. A computer-administered health screening interview for hospital personnel. MD Comput. 1995 Jan-Feb;12(1):25-30. PMID 7854075
- [Background] Bleich HL, Beckley RF, Horowitz GL, Jackson JD, Moody ES, Franklin C, Goodman SR, McKay MW, Pope RA, Walden T, et al. Clinical computing in a teaching hospital. N Engl J Med. 1985 Mar 21;312(12):756-64. doi: 10.1056/NEJM198503213121205. PMID 3838364
- [Background] Slack WV, Bleich HL. The CCC system in two teaching hospitals: a progress report. Int J Med Inform. 1999 Jun;54(3):183-96. doi: 10.1016/s1386-5056(99)00006-4. PMID 10405878
- [Background] Weizenbaum JE. ELIZA: a computer program for the study of natural language communication between man and machine. Commun Assoc Comput Mach 1966; 9: 36-45.
- [Background] Colby KM, Watt JB, Gilbert JP. A computer method of psychotherapy: preliminary communication. J Nerv Ment Dis. 1966 Feb;142(2):148-52. doi: 10.1097/00005053-196602000-00005. No abstract available. PMID 5936301
- [Background] Slack WV, Slack CW. Patient-computer dialogue. N Engl J Med. 1972 Jun 15;286(24):1304-9. doi: 10.1056/NEJM197206152862408. No abstract available. PMID 5024461
- [Background] Slack WV, Slack CW. Talking to a computer about emotional problems: a comparative study. Psychotherapy: Theory, Research, and Practice 1977; 14: 156-64.
- [Background] Slack WV, Porter D, Balkin P, Kowaloff HB, Slack CW. Computer-assisted soliloquy as an approach to psychotherapy. MD Comput. 1990 Jan-Feb;7(1):37-42, 58. PMID 2308504
- [Background] Starkweather JA. Computest: a computer language for individual testing, instruction, and interviewing. Psychol Rep. 1965 Aug;17(1):227-37. doi: 10.2466/pr0.1965.17.1.227. No abstract available. PMID 5826481
- [Background] Swedlow DB, Barnett GO, Grossman JH, Souder DE. A simple programming system ("driver") for the creation and execution of an automated medical history. Comput Biomed Res. 1972 Feb;5(1):90-8. doi: 10.1016/0010-4809(72)90010-9. No abstract available. PMID 5019502
- [Background] Angle HV, Carroll JA. Computer interview language: programming the on line interactive computer. Behav Res Meth Instrumentation 1979; 11: 379-83.
- [Background] Safran C, Rury C, Rind DM, Taylor WC. A computer-based outpatient medical record for a teaching hospital. MD Comput. 1991 Sep-Oct;8(5):291-9. PMID 1749339
- [Background] Horowitz GL, Bleich HL. PaperChase: a computer program to search the medical literature. N Engl J Med. 1981 Oct 15;305(16):924-30. doi: 10.1056/NEJM198110153051605. PMID 7024808
- [Background] Safran C, Herrmann F, Rind D, Kowaloff HB, Bleich HL, Slack WV. Computer-based support for clinical decision making. MD Comput. 1990 Sep-Oct;7(5):319-22. PMID 2243548
- [Background] Sands DZ, Halamka JD. PatientSite: patient centered communication, services, and access to information. In: Nelson R, Martin E, Safran C, eds. Consumer Informatics in a cyberhealth world. New York: Springer Verlag, scheduled for publication in 2003.
- [Background] Streiner DL, Norman GR. Health measurement scales: a practical guide to their development and use (second edition). Oxford: Oxford University Press, 1995.
- [Background] Fowler FJ. Improving survey questions: design and evaluation (Applied Social Research Methods Series Volume 38). London: SAGE Publications, 1995.
- [Background] Slack W. Computer-based interviewing system dealing with nonverbal behavior as well as keyboard responses. Science. 1971 Jan 8;171(3966):84-7. doi: 10.1126/science.171.3966.84. PMID 5538704
- [Background] Lucas RW. Computer interrogation: investigation of patients' response times. Int Res Commun Systems J Med Sci 1974; 2: 1176.
- [Background] Slack WV, Leviton A, Bennett SE, Fleischmann KH, Lawrence RS. Relation between age, education, and time to respond to questions in a computer-based medical interview. Comput Biomed Res. 1988 Feb;21(1):78-84. doi: 10.1016/0010-4809(88)90044-4. PMID 3345654
- [Background] Hays RD, Shaul JA, Williams VS, Lubalin JS, Harris-Kojetin LD, Sweeny SF, Cleary PD. Psychometric properties of the CAHPS 1.0 survey measures. Consumer Assessment of Health Plans Study. Med Care. 1999 Mar;37(3 Suppl):MS22-31. doi: 10.1097/00005650-199903001-00003. PMID 10098556
- [Background] Safran C, Rind D, Citroen M, Bakker AR, Slack WV, Bleich HL. Protection of confidentiality in the computer-based patient record. MD Comput. 1995 May-Jun;12(3):189-92. No abstract available. PMID 11644706
- [Background] Slack WV. The issue of privacy. MD Comput. 1997 Jan-Feb;14(1):8-11. No abstract available. PMID 9000843
- [Background] Slack WV. Private information in the hands of strangers. MD Comput. 1997 Mar-Apr;14(2):83-6. No abstract available. PMID 9066242
- [Background] Safran C, Porter D, Lightfoot J, Rury CD, Underhill LH, Bleich HL, Slack WV. ClinQuery: a system for online searching of data in a teaching hospital. Ann Intern Med. 1989 Nov 1;111(9):751-6. doi: 10.7326/0003-4819-111-9-751. PMID 2802433
- [Background] Slee VN, Slee DA, Schmidt HJ. Slee's health care terms (fourth edition). Saint Paul: Tringa Press, 2001.
- [Background] CLARK WA, MOLNAR CE. THE LINC: A DESCRIPTION OF THE LABORATORY INSTRUMENT COMPUTER. Ann N Y Acad Sci. 1964 Jul 31;115:653-68. No abstract available. PMID 14214042
- [Background] Slack WV, Kowaloff HB, Davis RB, Delbanco T, Locke SE, Safran C, Bleich HL. Evaluation of computer-based medical histories taken by patients at home. J Am Med Inform Assoc. 2012 Jul-Aug;19(4):545-8. doi: 10.1136/amiajnl-2011-000580. Epub 2012 Jan 11. PMID 22237866
- [Result] Slack WV, Kowaloff HB, Davis RB, Delbanco T, Locke SE, Bleich HL. Test-retest reliability in a computer-based medical history. J Am Med Inform Assoc. 2011 Jan-Feb;18(1):73-6. doi: 10.1136/jamia.2010.005983. Epub 2010 Nov 27. PMID 21113077
- See also: Beth Israel Deaconess Medical Center — http://www.bidmc.harvard.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited patients from the Healthcare Associates (HCA)and the Affiliated Physicians Group (APG) clinics of Beth Israel Deaconess Medical Center who were to see their primary care physician for the first time.
Pre-assignment Details: Forty-five patients enrolled in the Computer-based medical history study. Forty of these patients started the medical history and 32 of these patients completed the program.
Groups:
- Computer-based Medical History: The intervention is a computer-based medical history designed for patients to take in their homes via the Internet. The history is divided into 24 modules- family history, social history, cardiac history, pulmonary history, and the like. So far as possible, it is designed to model the comprehensive, inclusive, general medical history traditionally taken, when time permits, by a primary care doctor seeing a patient for the first time. It contains 232 primary questions asked of all patients about the presence or absence of medical problems. Of these, 215 have the preformatted mutually exclusive responses
Period: Overall Study
Arm/Group | Computer-based Medical History
Started | 40
Completed | 32
Not Completed | 8
Not completed — Withdrawal by Subject | 8

BASELINE CHARACTERISTICS:
Groups:
- Experimental: The intervention is a computer-based medical interview, which contains 232 primary questions that are asked of all respondents, and over 6000 frames (questions, explanations, suggestions, recommendations, and words of encouragement) that are available for presentation as determined by the patient's responses and the branching logic of the program.
Arm/Group | Experimental
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 36
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 18

OUTCOME MEASURES:

1. Primary Outcome: Patient Post Medical History Assessment Questionnaire
Description: The questionnaire consisted of 10 Likert scales questions assessing the computer-based history. The Likert scale ranged from 1 for 'Not at all' to 10 for 'Very'.
  We computed the mean of the responses to the question "How helpful were the questions when thinking about your health?" We also calculated a total score by averaging the mean scores of the 10 questions.
Time Frame: Immediately after taking the medical history
Population: We analyzed post medical history questionnaire responses for the 32 patients who completed the medical history patients.
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Computer-based Medical History: A computer-based medical history to take in their homes via the Internet. The history is divided into 24 modules- family history, social history, cardiac history, pulmonary history, and the like.
Arm/Group | Computer-based Medical History
Number analyzed (Participants) | 32
units on a scale
  Helpfulness questions thinking about health | 8.4 [4 to 10]
  Combined mean score for all 10 questions | 8.3 [6.7 to 9.3]

2. Primary Outcome: Patient Post Visit Questionnaire
Description: The questionnaire consisted of 6 Likert scales questions assessing helpfulness of the computer-based history for the patient at the time of the visit. The Likert scale ranged from 1 for 'Not at all helpful' to 10 for 'Very helpful'. We computed the mean of the responses to the question "How helpful was it for you to have taken the computer interview before seeing your doctor?" We also calculated a total score by averaging the mean scores of the 6 questions. In addition we calculated the combined mean of the responses of three of the patients whose doctors did not complete their post-visit questionnaire.
Time Frame: One day after the visit with the physician
Population: We analyzed post medical history questionnaire responses for the 23 patients who completed the medical history patients.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Computer-based Medical History
Number analyzed (Participants) | 23
units on a scale
  Helpfulness computer interview before visit | 8.3 [5 to 10]
  Combined mean for all 6 questions | 7.8 [7.4 to 8.4]
  Combined mean when 3 pts but not MDs entered data | 5.9 [5.0 to 7.0]

3. Primary Outcome: Physician Post Visit Questionnaire
Description: The questionnaire consisted of 6 Likert scales questions assessing helpfulness of the computer-based history for the physician at the time of the patient visit. The Likert scale ranged from 1 for 'Not at all helpful' to 10 for 'Very helpful'. We computed the mean of the responses to the questions "How helpful was it for your patient to have taken the computer interview before seeing you?" " and the question "To what extent do you think the computer summary helped you to provide better care to your patient?" We also calculated a total score by averaging the mean scores of the 6 questions. In addition we calculated the combined mean of the physician responses to the post-visit questionnaires when physicians filled out the questionnaire but their patients did not.
Time Frame: One day after the patient visit
Population: We analyzed post visit physician questionnaire responses for the patients who completed the medical history and who showed up for their appointment.
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Computer-based Medical History: The intervention is a computer-based medical history designed for patients to take in their homes via the Internet. The history is divided into 24 modules- family history, social history, cardiac history, pulmonary history, and the like. So far as possible, it is designed to model the comprehensive, inclusive, general medical history traditionally taken, when time permits, by a primary care doctor seeing a patient for the first time. It contains 232 primary questions asked of all patients about the presence or absence of medical problems. Of these, 215 have the preformatted mutually exclusive responses "Yes," "No," "Uncertain (Don't Know, Maybe)," "Don't understand," and "I'd rather not answer;" 10 have other sets of multiple choices, one response permitted; five have multiple choices with more than one response permitted, and two have numerical responses. There are also 6000 questions, explanations and suggestions, available for presentation dependent upon the patient's responses,
Arm/Group | Computer-based Medical History
Number analyzed (Participants) | 23
units on a scale
  Helpfulness pt taking computer hx before visit | 7.7 [5 to 10]
  How helpful was summary in providing care | 7.5 [4 to 10]
  Combined mean of all 6 questions | 7.6 [7.5 to 7.7]
  Combined mean MD's but not pts entered data | 7.2 [6.7 to 7.3]

4. Secondary Outcome: Number of Office Visits by Patients
Description: The experimental design was revised from a two arm experimental and control study to a one arm experimental study. Therefore this secondary measure no longer applied.
Arm/Group | Computer-based Medical History
Number analyzed (Participants) | 0

5. Secondary Outcome: Time Per Visit
Description: as for outcome 4
Arm/Group | Computer-based Medical History
Number analyzed (Participants) | 0

6. Secondary Outcome: Number of Telephone Calls and E-mail Messages Between Patients and Physicians
Description: as for outcome 4
Arm/Group | Computer-based Medical History
Number analyzed (Participants) | 0

7. Secondary Outcome: Completeness of Patients' Problem Lists
Description: as for outcome 4
Arm/Group | Computer-based Medical History
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Adverse Events were not collected/assessed for this study
Arm/Group | Computer-based Medical History
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes